CLINICAL TRIAL: NCT02555761
Title: Evaluation of the Safety and Effectiveness of Lastacaft® Ophthalmic Solution 0.25% (Alcaftadine) for the Prevention of Itching Associated With Allergic Conjunctivitis: A Postmarketing Surveillance Study in Korea
Brief Title: Safety and Efficacy of Lastacaft® for the Prevention of Itching Associated With Allergic Conjunctivitis in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 229666-007
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — alcaftadine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lastacaft®: One drop of Lastacaft® Ophthalmic Solution 0.25% (Alcaftadine) in each eye daily as prescribed as standard of care in clinical practice.
  Interventions: Drug: Alcaftadine Ophthalmic Solution 0.25%

INTERVENTIONS:
Drug: Alcaftadine Ophthalmic Solution 0.25% — Alcaftadine Ophthalmic Solution 0.25% (Lastacaft®) as prescribed as standard of care in clinical practice.
  Other Names: Lastacaft®

SUMMARY:
This post-marketing surveillance study will assess the safety and efficacy of Lastacaft® Opthalmic Solution 0.25% (Alcaftadine) for the prevention of itching associated with Allergic Conjunctivitis as prescribed as standard of care in clinical practice in Korea.

ELIGIBILITY:
Inclusion Criteria:

-Patients with itching associated with allergic conjunctivitis.

Exclusion Criteria:

-Patients with hypersensitivity to Lastacaft® or its components.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with itching associated with Allergic Conjunctivitis prescribed Lastacaft® as standard of care in clinical practice.
Sampling Method: Probability Sample
Enrollment: 3423 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bai, Study Director — Allergan
Locations (78):
- South Korea (78):
  - Seo-myeon St.Mary's Hospital, Busan
  - SeoMyeon St. Eye Clinic, Busan
  - Inje University Busan Paik Hospital, Busan
  - Soojung Eye Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Saint Mary Bright Eye Clinic, Busan
  - Daeyeon St.mary's Eye Center, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Pusan National University Yangsan Hospital, Busan
  - Barun Sungmo Eye Clinic, Busan
  - chamjoeun Ophthalmic Clinic, Busan
  - Soonchunhyang University Cheonan Hospital, Chungcheongnam-do
  - Cheil eye hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyoungpook national university hospital, Daegu
  - Daegu Nune Eye Hospital, Daegu
  - Saebom Eye Clinic, Daejeon
  - Jungbuwoorieye Clinic, Daejeon
  - Chonnam National University Hospital, Daejeon
  - Clean Eye clinic, Daejeon
  - Eye Love Eye Center, Daejeon
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hospital, Daejoen
  - Konyang University Hospital, Daejoen
  - St. Mary's Eye center, Geyonggi-do
  - Eins Eye Clinic, Geyonsangnam-do
  - Happ Eye 21, Gwangju
  - Gwang Ju Eye Clinic, Gwangju
  - Bora Eye Clinic, Gwangju
  - Myongji Hospital, Gyeonggi-do
  - Munsan Jeil Eye Clinic, Gyeonggi-do
  - Seoul Shinsegae Eye Center, Gyeonggi-do
  - Eagle Eye Center, Gyeonggi-do
  - Anyang Seoul Eye Clinic, Gyeonggi-do
  - Noon-Sarang Eye Hospital, Gyeonggi-do
  - Bright eye, Gyeonggi-do
  - Ansan Yonsei Eye Center, Gyeonggi-do
  - Yonsei Dream Eye Clinic, Gyeonggi-do
  - Bright Kim's Eye Clinic, Gyeongsangnam-do
  - Fatima ophthalmology, Gyeongsangnam-do
  - Gowoon eye clinic, Gyeongsangnam-do
  - Sungmo Eye Hospital, Haeundae-gu
  - Hangil Eye Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Renessance eye center, Incheon
  - Bupyung ST.Mary's eye clinic, Incheon
  - Pureun Eye Center, Jeollabuk-do
  - Onuri Eye Hospital, Jeollabuk-do
  - Seoul Eye Clinic, Jeollanam-do
  - National Health Insurance Service Ilsan Hospital, Kyounggi-do
  - Yonsei Woori Eye Clinic, Seoul
  - Gangnam ST. Mary's Eye Center, Seoul
  - Hplus Eye Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Saevit Eye Center, Seoul
  - Sinchon Yeonsei Eye Hospital, Seoul
  - Central seoul eye center, Seoul
  - Ian Eye Center, Seoul
  - Lee, Im-sun Eye Clinic, Seoul
  - Yonsei Eye Clinic, Seoul
  - Asan Medical Center, Seoul
  - See Samsung Eye Center, Seoul
  - Yoon Ho Eye Hospital, Seoul
  - Apgujeong Eye Center, Seoul
  - Joeunnun Vision Clinic, Seoul
  - Nune Eye Hospital, Seoul
  - GS eye clinic, Seoul
  - Lee Eye Institute, Seoul
  - Samsung medical center, Seoul
  - The catholic university of korea Seoul ST. Mary's Hospital, Seoul
  - Su Yonsei Eye Clinic, Seoul
  - Kim's Eye Hospital, Seoul
  - Bright Seoul Ophthalmology, Seoul
  - The Catholic Unoveristy of Korea, Seoul St Mary's Hospital, Seoul
  - Severance Hospital, Seoul
  - Park Chang Soo Eye Clinic, Seoul

REFERENCES:
- See also: More Information — http://allerganclinicaltrials.com